CLINICAL TRIAL: NCT04157400
Title: Neuromodulation of Motor and Sensory Spinal Pathways in Subjects Undergoing Epidural Spinal Cord Stimulation
Brief Title: Effect of Epidural Stimulation on Muscle Activation and Sensory Perception
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Nathan Rowland, Assistant Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00089881
Record Dates: First submitted 2019-11-04; First posted 2019-11-08 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-01

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Epidural Spinal Cord Stimulation (Experimental): Subjects with chronic pain that have been scheduled to receive spinal cord simulators for standard of care treatment.
  Interventions: Device: Intraoperative Parameter Testing; Device: Proprioception Testing During Stimulation; Device: Gait Analysis During Stimulation

INTERVENTIONS:
Device: Intraoperative Parameter Testing — Step 1: Recording and stimulation of spinal potentials during insertion of epidural spinal stimulator paddle
  Once the epidural paddle is placed, study procedures will begin by connecting the terminals of the paddle to an electrophysiological recording device for signal amplification and filtering. Using this recording setup, motor evoked potential (MEP) and somatosensory evoked potential (SSEP) protocols will be performed to determine motor and sensory thresholds, respectively. Next, the surgical procedure will resume and after the implantable pulse generator (IPG) has been placed, study procedures will begin again and include activation of both low-frequency tonic stimulation (LFTS) and high-frequency burst stimulation (HFBS) patterns from the inserted paddle while recording EMG signals.
Device: Proprioception Testing During Stimulation — Step 3: Proprioception testing
  The research team will investigate the perceived change in knee joint angle and direction of movement reported by the subject in a Threshold to Detect Passive Movement (TTDPM). The TTDPM protocol will begin with the subject sitting in the Biodex testing seat, with the non-tested leg hanging freely and the tested leg strapped to the rotating arm of the dynamometer at the lower shank. The subject will be blinded as to the mode and intensity of stimulation: HFBS, LFTS, or no stim. The TTDPM will consist of at least 10 trials for each stimulation condition chosen based on SCM outcomes. The subject has control of a kill-switch that immediately halts movement of the rotating arm, which is to be activated once the subject perceives movement OR if the subject begins to feel any pain or discomfort throughout the task.
Device: Gait Analysis During Stimulation — Step 4: Body weight support and treadmill (BWST) testing
  Similar to step 2, LFTS and HFBS patterns will be compared by systematically testing each individual contact on the paddle while investigating for changes in stepping speed, pattern and EMG moduling complexity. Regarding EMG module analysis, muscle activity will be recorded bilaterally via surface EMG from lower extremity musculature. Furthermore, subjects will also have active LED markers placed over their clothes in order to track whole body kinematics throughout this portion of the study.
  To optimize capture of steady state data on the treadmill, each subject will walk for approximately 10 sec prior to the 30 sec of data collection (40 sec per trial). This will allow capture of at least 10 consecutive steady state gait cycles (depending on cadence) per each amplitude selection for each stimulation delivery technique, which will be defined by parameters found during walking SCM.

SUMMARY:
Each year, an estimated 34,000 individuals undergo epidural spinal cord stimulation (SCS) surgery to address debilitating chronic low back and leg pain (CLBLP). Although the commercial application of SCS to treat CLBLP was approved by the FDA in 1989, only in the past decade have significant advancements in stimulator technology been introduced. For instance, traditional SCS devices achieved reduction in pain using a type of stimulation known as low-frequency tonic stimulation (LFTS, below 100 Hz), which was dependent on induction of paresthesias (i.e., a tingling sensation) over the areas of pain perception. However, investigators now know that LFTS compromises sensory information flowing back to the spinal cord, which can be important in other spinal cord functions such as proprioception and movement. On the other hand, recent innovations in stimulator technology now provide the capability to apply stimulation frequencies up to 10,000 Hz along with complex waveform patterns - known as high frequency burst stimulation or HFBS - that can mitigate pain perception without the induction of paresthesias and the negative consequences on proprioception and movement. We propose to study the effects of these recently introduced features in SCS technology on motor and sensory spinal thresholds, proprioception and movement in subjects with CLBLP.

The spinal cord relies on input from the motor cortex and surrounding extremities to initiate specific muscle recruitment, and recent evidence suggests that preservation of temporally specific proprioceptive information via dorsal column primary afferent fibers is critical for natural motor behaviors such as ambulation. Since the spinal cord is exposed during the placement of the SCS device, information about a subject's motor and sensory spinal pathways can be easily obtained during the regular course of the procedure and compared to proprioceptive and motor responses once the subject is awake and moving with the device turned on. Our lab specializes in electrophysiological recordings in subjects undergoing spinal cord stimulator (SCS) implantation for CLBLP, while MUSC's Locomotion Laboratory specializes in quantifying proprioception and movement in human subjects. In this proposal, investigators will apply these techniques to subjects with CLBLP to determine effects of spinal neuromodulation on motor and sensory thresholds, proprioception, and kinematics.

DETAILED DESCRIPTION:
Definitions and nomenclature:

Spinal cord stimulation (SCS) will be performed using a 32-electrode paddle array implanted in the dorsal epidural space along the thoracolumbar region of the spinal cord. The array will be powered by a multiple independent current-controlled (MICC) implantable pulse generator (IPG) connected to the paddle per standard of care procedures for SCS implantation. In addition, as per standard of care, motor evoked potential (MEP), somatosensory evoked potential (SSEP) and electromyography (EMG) will be performed via the IOMAX intraoperative neuromonitoring system. The SCS system will be placed for clinical purposes, i.e., treatment of chronic pain, however, the investigators will collect data at various points during the placement. The study procedures will add 15 minutes to the surgery. MUSC's Locomotion Rehabilitation Laboratory - located at the College of Health Professions Building C - houses a Biodex Pro System 4 isokinetic/isometric dynamometer. The Biodex will standardize application of passive isokinetic knee flexion/extension trials to each blinded subject for proprioceptive investigations, which will be referred to as threshold to detect passive movement (TTDPM) throughout the rest of this document. Finally, MUSC's Locomotor Energetics and Assessment Laboratory - also located at the College of Health Professions Building C - houses a dual belt Instrumental Treadmill that is coplanar with the floor and will be used during all walking events. The laboratory also has a 12-camera motion capture system that utilizes active infrared LED tracers to track kinematic positioning data and will be used during all walking events. Another tool offered by the lab is a 16-channel EMG system which utilizes surface electrodes to detect target muscle activity and will also be used during all walking events. In all, expected total duration of the study to be approximately 30 days.

Device use:

The epidural stimulator paddle and IPG are FDA-approved, commercially available devices designed to treat chronic pain of the back and lower extremities and will be used for their intended clinical purpose - electrical stimulation of dorsal column fibers to mitigate pain perception. The research use of this device, which will add approximately 15 minutes to the surgery, involves recording/stimulating from the device during the standard of care intraoperative neuromonitoring protocol. Regardless of study participation, the stimulator paddle and IPG will be implanted according to standard of care for the pre-planned SCS surgery. The IOMAX intraoperative neuromonitoring system, equipment owned by MUSC and operated by MUSC neurophysiology staff, is a commercially available device used during standard of care spinal surgical procedures, such as SCS implantation. Regardless of study participation, intraoperative neuromonitoring via IOMAX will take place according to standard of care for the pre-planned SCS surgery. The following devices are used for research purposes only. The Biodex Pro System 4, used regularly by physical rehabilitation researchers here at MUSC, is a commercially available device that will be used solely as a research tool to deliver passive isokinetic knee flexion/extension during the TTDPM. The Instrumental Treadmill, GAITRite mat, motion capture system, and MA300 EMG system are all commercially available devices that are used by MUSC researchers at the College of Health Professions to perform extensive gait analysis in subjects with various neurological deficits. Gait analysis is being performed for research purposes only, and is not standard of care for patients receiving SCS surgery.

Number of Subjects:

Investigators propose to study 5 individuals with CLBLP. A prior study conducted by Formento et al, 2018 using SCS and proprioceptive testing published a standard error and 95% confidence interval using successful and unsuccessful SCS trial attempts (p < 0.05 among LFTS parameters and no stimulation, with a minimum of 10 trials per stimulation setting.) Based on this, investigators expect that a small population will exhibit similar variance. The subject sample size is in direct comparison to sample sizes of previous proof of concept studies regarding SCS for spinal cord physiology biomarker sampling. The research team plans to use a two-way repeated measures ANOVA model in order to investigate the varying differences in stimulation type and kinematic parameters. A Post hoc comparison will be made using a Tukey adjustment.

Recruitment Methods:

During the subject's preoperative clinic visit, the PI will ask the potential participant if they would like to learn more about the study. If so, the PI will introduce the study and ask if he can answer any further questions about the study before inviting in the PI's physician assistant (listed as a study team member). If not, the PI will leave the room and the PI's physician assistant will review a prescreening checklist to determine whether subjects may be eligible for the study (no information obtained during the prescreening will be documented as research data). Potential participants will be asked to confirm that they are between the ages of 18 and 80, that they have been previously diagnosed with CLBLP by a pain specialist, whether they feel they cannot provide research consent physically and/or cognitively, and whether they have any prior history of spinal neoplasm, infection, arteriovenous malformation and/or radiation to the spine. If potential participants answer no to either of the first two questions or yes to either of the remaining questions, they will be considered ineligible for the study.

Careful attention will be placed on good communication. It will be emphasized that participation in the study is not necessary for standard of care medical treatment for their condition. It will also be emphasized that the subject can withdraw from the study at any time.

Data Management:

Once a potential participant is asked if they would like to learn more about the study, they will be assigned a participant ID. Participant IDs will be assigned consecutively. Investigators will maintain a database that accurately reflects all potential subjects that were approached about the study and the results of eligibility evaluation. For eligible subjects, the specific types of data that will be collected include: 1) analog local field potentials from the SCS, MEP, SSEP and EMG electrodes, 2) digital and analog output signals from the IOMAX intraoperative neuromonitoring device, 3) digital, time-stamped, physical displacement data captured from the Biodex machine, 3) digital, time-stamped, positioning data produced by the PhaseSpace software, 5) videography data, and 6) any available imaging data (dicom files). Raw data will remain on lab-owned data acquisition machines with encrypted hard drives and stored behind a locked door when not directly supervised. Data will be copied from all lab-owned data acquisition machines and/or hospital-owned data servers to a password protected network server accessible from the lab under the IRB protocol number and participant ID. This will constitute the master copy of all data for the lab and will consist of separately stored coded and identifiable folders. The purpose of keeping a copy of the raw data is in case the server is interrupted, and it is necessary to reconstruct the data. Portions of data will be copied to end-user devices (e.g., desktop, laptop, etc) for data analysis, however only the portion needed for analysis will be copied. Any end-user device such as a laptop that physically leaves the lab will be encrypted with MUSC-approved software which uses the AES encryption algorithm in cipher block chaining or XTS mode with a 256-bit key. Desktop machines used for analysis that do not leave the lab and are stored in a locked laboratory will not be encrypted. All data on data acquisition and end-user devices will be deleted at the conclusion of the study. No PHI will be stored on any data acquisition machine or end-user device. A linking database associating the participant ID and subject identifiers will be maintained on MUSC Box, separately from the research data. Subject identifiers to be collected include first and last name, gender, date of birth, social security number, medical record number, mailing address and telephone numbers. Telephone and medical record numbers are required for an approximate 7-day phone call made to subjects following SCS implantation. Additionally, investigators will collect information pertaining to disease severity for each subject, including Visual Analog Scale (VAS) scores, a common pain scale, and any other available rating scale scores. These measures will assist in correlating our physiological data with severity of disease for each subject. Videography data will be stored in the identifiable folder on the password protected network server. The purpose of this data is to correlate movement dynamics with physiology data. Finally, investigators will save imaging data on a password protected network server in order to analyze and correlate with the collected physiological data. Only IRB-approved personnel will have access to the linking database. Consent forms will be stored in a locked cabinet in a locked laboratory in the Clinical Sciences Building at MUSC.

Risks to Subjects:

All procedures will follow standard of care guidelines. Research staff will follow up with each participant by phone approximately one week after the surgical procedure, and during the approximate 30-day return, to make sure the participants are not having any problems. Nevertheless, this study still poses certain risks as outlined in the following sections:

Surgical complication

Due to the 15 extra minutes added to the surgery, connection of the paddle terminals outside the surgical field, and extra personnel in the room, there is a slightly increased risk of surgical infection. The extra risk of infection due to the research protocol does not increase this risk beyond the 1-5% overall historical risk of complications from the SCS surgical procedure.

TTDPM

While testing for proprioception retention of the lower extremities, subjects may encounter discomfort due to non-volitional muscle activation that hinders passive movement. To mitigate this risk, the Biodex system has a subject-controlled trigger that immediately stops the dynamometer's passive motion and may be activated at any time a subject experiences discomfort of pain during the test.

Overground and Treadmill Walking

Subjects will be asked to walk on a pressure sensitive mat at self-selected walking speeds and on a treadmill at self-selected walking speeds with each scenario having the subject in an upper thoracic safety harness which is tethered to the ceiling for fall protection. Despite the aforementioned safety measures, there still exists a risk of loss of balance, fall and potential injury. The risk to subjects through these tasks do not exceed risks involved with general physical therapy settings and may result in mild muscle fatigue or discomfort that generally subsides within a few days. Subjects will be given ample rest time and may have additional rest time at any point throughout data collection periods. Furthermore, subjects will be assisted during large movements or during potential transfers across different surfaces by an IRB-approved study member.

Photography and videography

Subjects will be videotaped during performance of supine / walking SCM and EMG moduling protocols. Investigators will also photograph and/or videotape any other aspect of the subject's research participation that will help investigators correlate the subject's condition with the EMG and kinematic data. The videos and photos recorded can include the full face, upper body, arms, and legs. Photography and videography carry a risk of loss of privacy. Photos and videos will be stored on a secure server. Only approved study personnel will have access to these files.

Loss of Confidentiality

Additional risks include loss of confidentiality. To mitigate this risk, a linking database associating the participant ID and subject identifiers will be maintained separately from the research data on a password protected server and only IRB-approved personnel will have access to the linking database.

ELIGIBILITY:
Research Inclusion Criteria

* Subjects diagnosed with CLBLP by a pain specialist with a documented referral for evaluation of SCS surgery by the pain specialist
* Subjects with the ability to walk
* Age 18-80

Research Exclusion Criteria

* Subjects with the inability to consent for themselves.
* Prior history of spinal neoplasm, infection, arteriovenous malformation and/or radiation to the spine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Rowland, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Potential participants will be informed during the consent process that information about them (including identifiable private information) may have all of their identifiers removed and used for future research studies or distributed to other researchers for future research without additional informed consent from them.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Not yet determined
Access Criteria: Not yet determined

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Spinal Cord Stimulation: Subjects with chronic pain that have been scheduled to receive spinal cord simulators for standard of care treatment.
  Intraoperative Parameter Testing: Step 1: Recording and stimulation of spinal potentials during insertion of epidural spinal stimulator paddle
Period: Overall Study
Arm/Group | Epidural Spinal Cord Stimulation
Started | 5
Completed | 1
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Epidural Spinal Cord Stimulation: Subjects with chronic pain that have been scheduled to receive spinal cord simulators for standard of care treatment.
  Intraoperative Parameter Testing: Step 1: Recording and stimulation of spinal potentials during insertion of epidural spinal stimulator paddle
  Once the epidural paddle is placed, study procedures will begin by connecting the terminals of the paddle to an electrophysiological recording device for signal amplification and filtering. Using this recording setup, motor evoked potential (MEP) and somatosensory evoked potential (SSEP) protocols will be performed to determine motor and sensory thresholds, respectively. Next, the surgical procedure will resume and after the implantable pulse generator (IPG) has been placed, study procedures will begin again and include activation of both low-frequency tonic stimulation (LFTS) and high-frequency burst stimulation (HFBS) patterns from the inserted paddle while recording EMG signals.
Arm/Group | Epidural Spinal Cord Stimulation
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Electromyography Response Amplitude
Description: During intraoperative testing of varying stimulation parameters, the research team plans to collect evoked potentials via electromyography (EMG) as the primary outcome for step one. Evoked potential amplitude, recorded at specific muscles of interest, will be collected for nerve root activation threshold. The research team plans to look at musculature receiving innervation from varying levels of the spinal cord in order to determine any difference among stimulation type regarding nerve root isolation.
Time Frame: Data collection for step one is expected to last approximately fifteen minutes during the spinal cord stimulation surgery.
Population: Three participants did not have sufficient data to analyze - 2 of the patients did not undergo the 2nd part of the protocol and 1 patient decided not to have surgery. One patient withdrew from the study prior to undergoing surgery.
Measure: Mean (Standard Error); unit: microvolts (mV)
Arm/Group | Epidural Spinal Cord Stimulation
Number analyzed (Participants) | 1
microvolts (mV)
  Vastus Lateralis (EMG); 40 Hz LFTS (Stimulation) | 33.7 (0.7)
  Vastus Lateralis (EMG); 600 Hz HFBS, 40 Hz interburst (Stimulation) | 122.1 (2.5)
  Tibialis Anterior (EMG); 40 Hz LFTS (Stimulation) | 39.2 (0.8)
  Tibialis Anterior (EMG); 600 Hz HFBS, 40 Hz interburst (Stimulation) | 69.7 (0.9)
  Soleus (EMG); 40 Hz LFTS (Stimulation) | 90.4 (1.2)
  Soleus (EMG); 600 Hz HFBS, 40 Hz interburst (Stimulation) | 143.0 (2.6)
Statistical Analysis 1: Comparison: Epidural Spinal Cord Stimulation; Test type: Other; p < 0.01, Kruskal-Wallis

2. Primary Outcome: Proprioception Testing
Description: Proprioception signaling will be tested using a Biodex machine that can apply passive flexion/extension at the knee while the subject reports 1) Feeling of movement and 2) Direction of movement. Specific data of interest will be the amount of degrees of flexion/extension of the knee that have occurred before the subject perceives the movement, which is reflective of proprioceptive signaling. Testing while experiencing varying types of stimulation will yield important information regarding physiological sensory modulation from the stimulator. The research team plans to use a repeated measures two-way ANOVA with epidural stimulation type and current amplitude of above and below EMG activation threshold to investigate effects on proprioception detection signaling.
Time Frame: Data collection for step two is expected to last approximately two hours.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Degrees of Flexion / Extension
Arm/Group | Epidural Spinal Cord Stimulation
Number analyzed (Participants) | 1
Degrees of Flexion / Extension
  Degrees of passive knee flexion / extension before detection: No stimulation | 3.93 (0.35)
  Degrees of passive knee flexion / extension before detection: 40 Hz LFTS | 6.71 (0.63)
  Degrees of passive knee flexion / extension before detection: 600 Hz HFBS, 40 Hz interburst | 4.52 (0.21)
Statistical Analysis 1: Comparison: Epidural Spinal Cord Stimulation; Test type: Other; p < 0.001, ANOVA

3. Primary Outcome: Change in Electromyography Microvoltage Signal During Walking
Description: During gait analysis, the research team plans to collect surface electromyography (EMG) signals of lower extremity musculature to measure activation synergies and amplitudes. Segments of EMG that are recorded during walking will be analyzed with an algorithm that yields hierarchal complexities representing muscle synergies known as EMG moduling. The research team plans to use a two-way repeated measures ANOVA model in order to investigate the varying differences in stimulation type and effect on EMG module complexity to investigate the relationship between sensory pathway modulation and motor control during functional task.
Time Frame: Data collection for step three is expected to last approximately two hours.
Population: as for outcome 1
Measure: Number; unit: microvolts (mV)
Groups:
- Epidural Spinal Cord Stimulation: Subjects with chronic pain that have been scheduled to receive spinal cord simulators for standard of care treatment.
  .
Arm/Group | Epidural Spinal Cord Stimulation
Number analyzed (Participants) | 1
microvolts (mV)
  EMG Module Complexity During No Stimulation | 4.1
  EMG Module Complexity During 40 Hz LFTS | 2.6
  EMG Module Complexity During 600 Hz HFBS, 40 Hz interburst | 3.2
Statistical Analysis 1: Comparison: Epidural Spinal Cord Stimulation; Test type: Other; Segments of EMG recorded during walking at self-selected walking speed were used to investigate complexity of muscle synergies using a nonnegative matrix factorization (NNMF) algorithm (MATLAB®, Mathworks, Natick, MA). The approach involves calculation of an mxt matrix of the original EMG data (EMG0), where m represents the number of muscles being measured and t represents a time base normalized to percentage of gait cycle. The algorithm also calculates two surrogate matrices, mxn and nxt, where n is the amplitude of muscle activation. The product of the surrogate matrices are considered a reconstruction of EMG (EMGr). EMGr for each module is then compared to EMG0 by finding the variability accounted for (VAF). A threshold necessary for module classification was chosen to be 90% for all conditions (8 muscles + 6 phases of gait) based on similar studies in the literature. Classifications were not increased unless the higher module VAF was at least 5% higher than the preceding module

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse / Serious Adverse Event Questionnaire given at 7 day followup phone call and 30 day followup visit.
Arm/Group | Epidural Spinal Cord Stimulation
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-15): https://cdn.clinicaltrials.gov/large-docs/00/NCT04157400/Prot_SAP_001.pdf